CLINICAL TRIAL: NCT00954993
Title: A Multiple Dose Study to Evaluate Pharmacokinetics and Hepatitis C Virus RNA Following Administration of MK-7009 in Hepatitis C Infected Patients
Brief Title: Pharmacokinetics of Vaniprevir (MK-7009) and Hepatitis C Virus RNA Levels After Vaniprevir Treatment (MK-7009-029)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was stopped for business and program changes. At no time was the safety of any participants at risk.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7009-029; 2009-013076-41 (EudraCT Number)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C Virus (HCV); Vaniprevir; MK-7009
MeSH Terms: conditions — Hepatitis C | interventions — vaniprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaniprevir 600 mg - 300 mg (Experimental): For each participant in period 1, 600 mg of Vaniprevir was taken twice daily on Days 1-3 and a single dose of Vaniprevir 600 mg was taken on Day 4. Period 1 was followed by a minimum 30-day, up to approximately 140 day, washout interval. In period 2, 300 mg of Vaniprevir was taken twice daily by each participant on Days 1-3 and a single dose of Vaniprevir 300 mg was taken on Day 4.
  Interventions: Drug: Vaniprevir

INTERVENTIONS:
Drug: Vaniprevir — Period 1: Vaniprevir 600 mg twice daily on Days 1-3 and a single dose of Vaniprevir 600 mg on Day 4. Period 2: Vaniprevir 300 mg twice daily on Days 1-3 and a single dose of Vaniprevir 300 mg on Day 4. There was at least a 30-day (up to approximately 140-day) washout interval between periods 1 and 2.
  Other Names: MK-7009

SUMMARY:
This study will evaluate the hepatic (liver) and plasma pharmacokinetics of Vaniprevir (MK-7009) by evaluation of ribonucleic acid (RNA) of the hepatitis C virus (HCV) in genotype 1, HCV-infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female between 40 to 65 years of age at the prestudy (screening) visit
* Participant has a Body Mass Index (BMI) ≥18.5 kg/m2 and ≤36.0 kg/m2.
* Participant requires a diagnostic biopsy, per local treatment guidelines, to monitor progression of liver disease.
* Participant has chronic compensated, genotype 1 HCV infection as defined by positive serology for HCV and detectable HCV RNA in peripheral blood
* Participant met pre-specified criteria based on laboratory values at screening for the following: -- Alanine aminotransferase (ALT): ≤400 U/L -- Aspartate aminotransferase (AST): ≤400 U/L -- Total bilirubin: ≤2.4 mg/dL -- Direct bilirubin: ≤1.0 mg/dL -- Creatinine clearance (Clcr): ≥60 mL/min (by the Cockcroft-Gault equation*) -- Albumin: ≥3.3 g/dL -- Alkaline phosphatase: ≤260 U/L -- Hemoglobin: ≥13 g/dL (men), ≥12 g/dL (women) -- White blood cell count: 3.8 to 10.7 ×103/μL -- Absolute neutrophil count: ≥1.5 ×103/μL -- Platelet count: ≥120 ×103/μL -- International normalized ratio (INR): ≤1.2 -- Thyroid stimulating hormone (TSH): 0.34 to 5.60 μIU/mL -- Alpha fetoprotein (AFP): <100 ng/mL
* Participant does not have cirrhosis as confirmed by FibroSure™/FibroTest®
* Participant is treatment-experienced, with regard to prior treatment for chronic HCV infection
* Participant has the ability to avoid use of anticoagulants, nonsteroidal anti-inflammatory agents and aspirin for at least five (5) days preceding the initial liver biopsy and continuing throughout the entire study

Exclusion Criteria:

* Participant is under the age of legal consent, is mentally or legally incapacitated/ institutionalized, has significant emotional problems at the time of prestudy screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
* Participant has a history of stroke, chronic seizures, or major neurological disorder
* Participant did not achieve a viral response to prior treatment with licensed interferon-based therapy (i.e., is a 'null responder'). Viral response is defined by a >= 2-log^10 decline in HCV viral RNA within the first 12 weeks of therapy.
* Participant has previously been treated with an NS3/4A protease inhibitor for chronic HCV infection
* Evidence of high grade bridging fibrosis (eg, METAVIR score >3, Ishak score >4 or Scheuer score >3) from prior liver biopsy within 3 years of study entry
* Participant has evidence or history of chronic hepatitis not caused by HCV including but not limited to non-HCV viral hepatitis, nonalcoholic steatohepatitis (NASH), drug-induced hepatitis or autoimmune hepatitis. Note: Participants with history of acute non-HCV-related hepatitis which resolved >6 months before study entry can be enrolled.
* Participant has clinical or laboratory evidence of cirrhosis or other advanced liver disease
* Participant has decompensated liver disease as indicated by a history of ascites, hepatic encephalopathy, or bleeding esophageal varices
* Participant has been diagnosed or suspected of hepatocellular carcinoma
* Participant has coinfection with human immunodeficiency virus (HIV)
* Participant has positive Hepatitis B surface antigen or other evidence of active Hepatitis B infection
* Participant has a history of gastric bypass surgery, bowel resection or other disorder that in the opinion of the investigator may interfere with the absorption of the study medication
* Participant has a history of clinically significant uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Participant has a history of neoplastic disease (including leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment
* Participant consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL], wine [125 mL], or distilled spirits [25 mL]) per day
* Participant is currently a regular user (including use of any illicit drugs or has a history of drug (including alcohol) abuse within the last 3 months
* Female participant is pregnant, lactating, expecting to conceive or donate eggs, or is of childbearing potential and unwilling to commit to two methods of birth control as outlined in inclusion criterion
* Male Participant is planning to impregnate or provide sperm donation or has a female sexual partner of childbearing potential and is unwilling to commit to using two methods of birth control as outlined in inclusion criterion

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01-13 (Actual); Primary Completion 2011-03-04 (Actual); Study Completion 2011-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-029&kw=7009-029&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaniprevir 600 mg - 300 mg Arm: For each participant in period 1, 600 mg of Vaniprevir was taken twice daily on Days 1-3 and a single dose of Vaniprevir 600 mg was taken on Day 4. Period 1 was followed by a minimum 30-day, up to approximately 140 day, washout interval. In period 2, 300 mg of Vaniprevir was taken by each participant twice daily on Days 1-3 and a single dose of Vaniprevir 300 mg was taken on Day 4.
Period: Period 1
Arm/Group | Vaniprevir 600 mg - 300 mg Arm
Started | 3
Completed | 3
Not Completed | 0
Period: Washout
Arm/Group | Vaniprevir 600 mg - 300 mg Arm
Started | 3
Completed | 3
Not Completed | 0
Period: Period 2
Arm/Group | Vaniprevir 600 mg - 300 mg Arm
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vaniprevir 600 mg - 300 mg Arm
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) (0-12 Hrs) of Vaniprevir in the Liver
Description: Participants were treated with vaniprevir twice daily on days 1,2, and 3. On treatment Day 4 participants were treated once with vaniprevir; then core needle liver biopsies were to be collected at 6, 12 and 24 hours postdose to determine the AUC of vaniprevir. AUC is the integrated area under the curve for plasma concentration of vaniprevir over time.
Time Frame: 6, 12 and 24 hours postdose on day 4 of each period (up to Day 148)
Population: Since only a single liver sample timepoint at either 6 or 12 hours was obtained from each participant, and no 24 hour timepoint was collected from any participant due to the early termination of the study, the AUC (0-12 hrs) was not calculated
Groups:
- 600 mg Dose of Vaniprevir: 600 mg of Vaniprevir was taken twice daily on Days 1-3 of Period 1 and a single dose of Vaniprevir 600 mg was taken on Day 4 of Period 1.
- 300 mg Dose of Vaniprevir: 300 mg of Vaniprevir was taken twice daily on Days 1-3 of Period 2 and a single dose of Vaniprevir 300 mg was taken on Day 4 of Period 2.
Arm/Group | 600 mg Dose of Vaniprevir | 300 mg Dose of Vaniprevir
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Concentration of Vaniprevir in the Liver
Description: Participants were treated with vaniprevir on days, 1,2, and 3. On treatment Day 4 participants were treated once with vaniprevir; then core needle liver biopsies were collected at 6, 12, and 24 hours postdose to determine the concentration of vaniprevir in the liver.
Time Frame: 6, 12 and 24 hours postdose on day 4 of each period (up to day 148)
Population: Participants treated with vaniprevir who had a liver biopsy were analyzed as two separate groups that received 600 mg and 300 mg doses . No biopsies were collected at the 24 hour timepoint.
Measure: Median (Full Range); unit: nM
Arm/Group | 600 mg Dose of Vaniprevir | 300 mg Dose of Vaniprevir
Number analyzed (Participants) | 3 | 3
nM
  6 Hours (n=2) | 169000 [79100 to 258000] | 84600 [67500 to 102000]
  12 Hours (n=1) | 53700 [53700 to 53700] | 29400 [29400 to 29400]

3. Primary Outcome: Apparent Terminal Half-life (t-1/2) of Vaniprevir in the Liver
Description: Participants were treated with vaniprevir twice daily on days 1,2, and 3. On treatment Day 4 participants were treated once with vaniprevir; then core needle liver biopsies were to be collected at 6, 12 and 24 hours postdose to determine the t-1/2 of vaniprevir. The t-1/2 is the time taken to eliminate half the amount of vaniprevir.
Time Frame: 6, 12 and 24 hours postdose on day 4 of each period (up to day 148)
Population: Since only a single liver sample timepoint was obtained from each participant at either 6 or 12 hours, and the 24 hour timepoint was not collected from any participant due to the early termination of the study, the t-1/2 could not be determined.
Arm/Group | 600 mg Dose of Vaniprevir | 300 mg Dose of Vaniprevir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately Day 148
Arm/Group | 600 mg Dose of Vaniprevir | 300 mg Dose of Vaniprevir
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg Dose of Vaniprevir (N=3) | 300 mg Dose of Vaniprevir (N=3)
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anger (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.